CLINICAL TRIAL: NCT01991223
Title: Efficacy of Dexmedetomidine for the Therapy of Catheter-related Bladder Discomfort
Brief Title: Dexmedetomidine for Catheter-related Bladder Discomfort
Acronym: CRBDEX
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Hee-Pyoung Park, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CRBD_DEX_PHPKHC; CRBD_SNUH1 (Other Grant/Funding Number: Seoul National University of Hospital)
Record Dates: First submitted 2013-11-18; First posted 2013-11-25 (Estimated); Last update posted 2014-03-19 (Estimated); Status verified 2014-03

CONDITIONS: Pain; Blood Pressure; Nausea; Vomiting; Arrhythmia
MeSH Terms: conditions — Pain; Nausea; Vomiting; Arrhythmias, Cardiac

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo group (Placebo Comparator): NS infusion will be done during surgery.
  Interventions: Drug: NS infusion
- Dex group (Experimental): DEX infusion will be done during surgery.
  Interventions: Drug: Dex infusion

INTERVENTIONS:
Drug: Dex infusion — Dexmedetomidine will be injected (1 mcg/kg for 10 minutes and afterward 0.3 mcg/kg/hr)
  Arms: Dex group
Drug: NS infusion — Normal saline will be infused during surgery
  Arms: Placebo group

SUMMARY:
To evaluate the efficacy of dexmedetomidine for the prevention of catheter-related bladder discomfort

DETAILED DESCRIPTION:
After transurethral bladder resection, large-sized foley catheter have been used for drainage of urine and residual blood. Because of urinary catheterization, patients usually experiences catheter-related bladder discomfort defined as a burning sensation with an urge to void or discomfort in the supra-pubic region caused by catheter- related bladder irritation.

Dexmedetomidine is an alpha-2 antagonist and used as an analgesic agent. The investigators try to evaluate The efficacy of dexmedetomidine for the treatment of catheter-related bladder discomfort

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for transurethral bladder resection
* ASA I-III

Exclusion Criteria:

* Patient who disagrees to participate this investigation
* Patient with severe cardiovascular disease
* Patient with small-sized foley catheter (less than 18 Fr.)
* Patinets with any urinary tract obstructions
* Patient with hyperactive or neurogenic bladder
* Patients with chronic renal failure
* Patient with morbidly obese
* Patients with neurogenic disorder
* Patient with medications for chronic pain

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Estimated)
Dates: Start 2013-11; Primary Completion 2014-11 (Estimated); Study Completion 2014-11 (Estimated)

PRIMARY OUTCOMES:
The number of patients with catheter-related bladder discomfort | at postoperative 1 hour
  catheter-related bladder discomfort at postoperative 1 hour was evaluated as none, mild, moderate, severe. The number of patients with mild, moderate, severe discomfort will be calculated and compared between groups.

SECONDARY OUTCOMES:
Catheter-related bladder discomfort | at postoperative 0, 1, 6, 24 hours
  Catheter-related bladder discomfort will be evaluated as none, mild, moderate, severe at postoperative 0, 1, 6, 24 hours.
Pain at suprapubic area | at postoperative 0, 1, 6, 24 hours
  Pain at suprapubic area will be evaluated using NRS (0:none, 100:worst imaginable) at postoperative 0, 1, 6, 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Hee-Pyoung Park, Principal Investigator — Seoul National University of Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Kim HC, Lee YH, Jeon YT, Hwang JW, Lim YJ, Park JE, Park HP. The effect of intraoperative dexmedetomidine on postoperative catheter-related bladder discomfort in patients undergoing transurethral bladder tumour resection: A double-blind randomised study. Eur J Anaesthesiol. 2015 Sep;32(9):596-601. doi: 10.1097/EJA.0000000000000196. PMID 25485879